CLINICAL TRIAL: NCT02513927
Title: The Effects of Nifedipine and Metoprolol on Blood Pressure Variability in Northern Chinese: a Randomized Crossover Study
Brief Title: The Effects of Nifedipine and Metoprolol on Blood Pressure Variability in Northern Chinese
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HT-2
Record Dates: First submitted 2015-07-21; First posted 2015-08-03 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
Keywords: Blood pressure variability; CCB; beta-receptor blockers; heart rate
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nifedipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): To observe the effects of metoprolol (95 mg) on blood pressure variation after 12 weeks of treatment.Then to observe the effects of Nifedipine (30 mg) on blood pressure variation after 12 weeks of treatment.
  Interventions: Drug: metoprolol; Drug: Nifedipine
- B (Active Comparator): To observe the effects of Nifedipine (30 mg) on blood pressure variation after 12 weeks of treatment. Then to observe the effects of metoprolol (95 mg) on blood pressure variation after 12 weeks of treatment.
  Interventions: Drug: metoprolol; Drug: Nifedipine

INTERVENTIONS:
Drug: metoprolol — Metoprolol was given orally in a dose of 95 mg/day to treat patients in the metoprolol group for 12 weeks.
Drug: Nifedipine — Nifedipine was given orally in a dose of 30 mg/day to treat patients in the amlodipine group for 12 weeks.

SUMMARY:
Hypertension is one of the most common cardiovascular diseases, which is a major risk factor for stroke and cardiovascular events. Traditionally, cardiovascular risk stratification in hypertensive patients was based on the average blood pressure (BP) measured in the clinic. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. Growing evidence demonstrated that BPV has considerable prognostic value for all-cause mortality and cardiovascular outcomes, independent of average BP.

At present, the normal range of BPV is not very clear. There are many studies about the effects of different kinds of drugs on blood pressure, but the clinical researches about the impacts of antihypertensive drugs on BPV are limited, and the conclusion is still controversial.

DETAILED DESCRIPTION:
Hypertension is one of the most common cardiovascular diseases, which is a major risk factor for stroke and cardiovascular events. Traditionally, cardiovascular risk stratification in hypertensive patients was based on the average blood pressure (BP) measured in the clinic. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. Growing evidence demonstrated that BPV has considerable prognostic value for all-cause mortality and cardiovascular outcomes, independent of average BP.

The hypertension prevalences in the high latitude and cold regions are much higher than those in the low latitude and warm regions. In China, the prevalences of hypertension are gradually increased from the South to the North. Heilongjiang province is the "high-risk" region for hypertension, with a prevalence of 30.48%. This may be due to the combined effects of lower average temperature and higher intake of salt and saturated fatty acid, which Increased sympathetic nerve excitability, and eventually lead to elevation of blood pressure. Therefore, it is essential to formulate the best treatment of hypertension according with the physical characteristics of northern Chinese.

At present, the normal range of BPV is not very clear. There are many studies about the effects of different kinds of drugs on blood pressure, but the clinical researches about the impacts of antihypertensive drugs on BPV are limited, and the conclusion is still controversial.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 75 included years old
* Postmenopausal women who are no more than 75 years older.
* Patients with essential mild to moderate uncomplicated hypertension (DBP<110mmHg and SBP<180mmHg measured with a validated automatic device in sitting position) after initiation or intensification of appropriate healthy lifestyle modification,
* Without antihypertensive treatment in 2 weeks.

Exclusion Criteria:

* History of cerebrovascular disease: ischemic stroke, cerebral haemorrhage and TIA.
* History of cardiovascular disease:unstable angina, myocardial infarction, coronary revascularization and congestive heart failure.
* History of renal impairment.
* History of Type I diabetes mellitus or Type II diabetes uncontrolled.
* History of liver impairment.
* History of alcoholism or drug abuse.
* Known symptomatic orthostatic hypotension.
* Contra-indications to treatment with investigate products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
24-hour Ambulatory Blood Pressure Monitoring | 3 years

SECONDARY OUTCOMES:
plasma uric acid level | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Twenty-four-hour ambulatory BP monitoring, Budapest, Budapest, Hungary